CLINICAL TRIAL: NCT02602327
Title: Phase I Study of Tas-102 and Radioembolization With 90Y Resin Microspheres for Chemo-refractory Colorectal Liver Metastases
Brief Title: Tas-102 and Radioembolization With 90Y Resin Microspheres for Chemo-refractory Colorectal Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Sirtex Medical (Industry); Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16452; NCI-2017-01321 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Colon Cancer; Rectal Cancer; Liver Metastases
Keywords: radioembolization; Yttrium-90; 90Y; Resin microspheres; Tas-102; Lonsurf; SIR-Sphere
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tas-102 and radioembolization (Experimental): Combination therapy with Tas-102 and radioembolization using 90Y resin microspheres
  Interventions: Drug: Tas-102; Device: SIR-Sphere

INTERVENTIONS:
Drug: Tas-102 — Oral nucleoside antitumor agent consisting of α,α,α-trifluorothymidine (FTD) and 5-chloro-6-(2-iminopyrrolidin-1-yl) methyl-2,4 (1H,3H)-pyrimidinedione hydro chloride (TPI) at a molar ratio of 1:0.5.
  Other Names: Lonsurf
Device: SIR-Sphere — 20-60mm resin microspheres containing Yttrium-90 (90Y, Y90) radioisotope
  Other Names: Yttrium-90 (Y90; 90Y) resin microspheres

SUMMARY:
This is a phase I dose escalation study (3+3 design) with a dose expansion arm (12 patients) designed to evaluate safety of the combination of Tas-102 and radioembolization using Yttrium-90 (90Y) resin microspheres for patients with chemotherapy-refractory liver-dominant chemotherapy-refractory metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
Randomized studies have demonstrated that Tas-102 has single agent activity against chemotherapy refractory colorectal cancer. A recent pre-clinical study has shown that Tas-102 may have activity as a radiation sensitizer in bladder cancer cell lines. Benefit of single agent Tas-102 against chemotherapy refractory colon cancer and the drug's promise a radiosensitizer make Tas-102 a potential candidate drug for testing in combination with radioembolization using Yttrium-90 resin microspheres in patients with liver-dominant chemotherapy-refractory mCRC. This is a phase I dose escalation study with a dose expansion arm designed to evaluate safety of the combination of Tas-102 and radioembolization using 90Y resin microspheres for patients with chemotherapy-refractory colon or rectal adenocarcinoma metastatic to the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older, and of any ethnic or racial group.
2. Diagnosis of unresectable metastatic colorectal adenocarcinoma with liver-dominant bilobar disease. Diagnosis may be made by histo- or cyto-pathology, or by clinical and imaging criteria.
3. Disease progression or intolerance to at least two prior Food and Drug Administration-approved therapeutic regimens.
4. If extrahepatic disease is present, it must be asymptomatic.
5. If a primary tumor is in place, it must be asymptomatic.
6. Measurable target tumors using standard imaging techniques (RECIST v. 1.1 criteria).
7. Tumor replacement < 50% of total liver volume.
8. Current Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 through screening to first treatment on study.
9. Completion of prior systemic therapy at least 14 days prior to enrollment.
10. Able to understand informed consent.

Exclusion Criteria:

1. At risk of hepatic or renal failure

   * Serum creatinine > 1.5 mg/dl
   * Serum bilirubin > 1.3 mg/ml
   * Albumin < 2.0 g/dL
   * Aspartate and/or alanine aminotransferase level > 5 times upper normal limit
   * Any history of hepatic encephalopathy
   * Cirrhosis or portal hypertension
   * Clinically evident ascites (trace ascites on imaging is acceptable)
2. Contraindications to angiography and selective visceral catheterization

   * Any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agents (e.g. closure device)
   * Severe allergy or intolerance to contrast agents, narcotics, or sedatives that cannot be managed medically
3. Symptomatic lung disease
4. Prior therapy with Tas-102.
5. Contraindications to Tas-102

   * Absolute neutrophil count < 1,500/μl
   * Platelet count < 75,000/μl
   * Allergy or intolerance to Tas-102
6. Unresolved toxicity of greater than or equal to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 2 due to prior therapies.
7. Evidence of potential delivery of

   * Greater than 30 Gy absorbed dose of radiation to the lungs during a single 90Y resin microsphere administration; or
   * Cumulative delivery of radiation to the lungs > 50 Gy over multiple treatments.
8. Evidence of any detectable Tc-99m macro aggregated albumin flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow.
9. Previous radiation therapy to the lungs and/or to the upper abdomen
10. Any prior arterial liver-directed therapy, including chemoembolization, bland embolization, and 90Y radioembolization
11. Any intervention for, or compromise of the ampulla of Vater
12. Active uncontrolled infection. Presence of latent or medication-controlled HIV and/or viral hepatitis is allowed.
13. Significant extrahepatic disease

    * Symptomatic extrahepatic disease (including primary tumor, if unresected).
    * Greater than 10 pulmonary nodules (each < 20 mm in diameter) or combined diameter of all pulmonary nodules > 15 cm.
    * Peritoneal carcinomatosis
14. Life expectancy less than 3 months
15. Pregnant or lactating female
16. In the investigator's judgment, any co-morbid disease or condition that would place the patient at undue risk and preclude safe use of radioembolization or Tas-102.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Determine dose limiting toxicities (DLT) | 56 days
  Any adverse events grade ≥ 3 will be reviewed by the treating interventional radiologist and medical oncologist within 24 hours of being informed event. If none of the 3 patients in a cohort experiences a DLT, another 3 patients will be treated at the next higher dose level. However, if 1 of the first 3 patients experiences a DLT, 3 more patients will be treated at the same dose level. The dose escalation will continue until at least 2 patients among a cohort of 3-6 patients experience DLTs (i.e., ≥ 33% of patients with a dose-limiting toxicity at that dose level) or until 3-6 patients had been treated at TAS-102 dose of 35mg/m2 per day in 2 divided doses (up to a maximum of 80 mg per dose) administered concurrently with radioembolization cycles 1 and 2 without experiencing a DLT. DLT window will be 56 days (cycle 1, day 1 to cycle 2, day 28). Dose limiting toxicity will be reached when one of the clinical and/or laboratory parameters are met
Maximum tolerated dose (MTD) | Up to 4 years
  Traditional 3+3 design will be used to determine the recommended dose for the dose expansion phase will be defined as the dose level just below this toxic dose level.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 4 years
  Radiographic overall response rate (measured in accordance to Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1) using imaging. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): 30% decrease in the sum of the longest diameter of target lesionsStable Disease (SD): Small changes that do not meet the criteria for CR, PR, or Progressive Disease (PD): 20% increase in the sum of the longest diameter of target lesions. ORR will be defined as a ratio of the number of patients who demonstrated complete response (CR) or partial response (PR) to the number of all evaluated patients.
Progression-free survival (PFS) | Up to 4 years
  PFS will be defined as a time period that started at enrollment, during which a patient neither progressed nor died based on radiographic response.
Hepatic progression-free survival (HPFS) | Up to 4 years
  HPFS will be defined as a time period that started at enrollment, during which a patient neither progressed in the liver nor died based on radiographic response.
Extrahepatic progression free survival (EHPFS) | Up to 4 years
  EHPFS will be defined as a time period that started at enrollment, during which a patient neither progressed outside the liver nor died based on radiographic response
Overall survival (OS) | Up to 12 months
  Overall Survival will be analyzed 12 months after the last patient is enrolled. Overall survival will be assessed using a two-sided, log-rank test. The survival function will be estimated using the Kaplan-Meier product limit method. In addition, two-sided 95% confidence intervals for the median overall survival will be computed
Biomarker response | Up to 4 years
  Proportion of patients with carcinoembryonic antigen (CEA) response with ≥ 50% decline from baseline (in patients with baseline level ≥ 3.2) post combination therapy with Tas-102 and 90Y radioembolization. Maximum percent change will be calculated. CEA level will only be followed for participants with elevated level (≥3.2) at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fidelman, MD, Principal Investigator — University of California, San Francisco; Katherine Van Loon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fidelman N, Atreya CE, Griffith M, Milloy MA, Carnevale J, Cinar P, Venook AP, Van Loon K. Phase I prospective trial of TAS-102 (trifluridine and tipiracil) and radioembolization with 90Y resin microspheres for chemo-refractory colorectal liver metastases. BMC Cancer. 2022 Dec 13;22(1):1307. doi: 10.1186/s12885-022-10401-0. PMID 36514060